CLINICAL TRIAL: NCT05464472
Title: Impact of Transcatheter Aortic Valve Implantation (TAVI) on Cognitive Functions
Acronym: KogniTa
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helios University Hospital Wuppertal (Other)
Responsible Party: Sponsor
Other Study IDs: Cardio 01
Record Dates: First submitted 2022-03-27; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Cognition Disorder
Keywords: Transcatheter Aortic Valve Implantation (TAVI); Cognitive Function; Aortic stenosis; Stroke; Frailty
MeSH Terms: conditions — Cognition Disorders; Aortic Valve Stenosis; Stroke; Frailty | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transcatheter Aortic Valve Implantation: Patients are assessed for cognitive function pre and post transcatheter aortic valve implantation.
  Interventions: Device: Transcatheter Aortic Valve Implantation (TAVI)
- Control matched population: Control matched population are assessed for cognitive function at day 0 and at 6 month

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation (TAVI) — Guideline/ FDA approved implantation of a Transcatheter Aortic Valve Implantation (TAVI)
  Groups: Transcatheter Aortic Valve Implantation

SUMMARY:
Interventional implantation of the aortic valve (Transcatheter Aortic Valve Implantation; TAVI) may alter neurocognitive functions. We aim to differentiate the changes in cognitive functions after a TAVI.

DETAILED DESCRIPTION:
Interventional implantation of the aortic valve (Transcatheter Aortic Valve Implantation; TAVI) is the treatment of choice for patients with symptomatic aortic valve stenosis >75 years with comorbidities. The reduction in complications and also in mortality after TAVI is due, among other things, to the constant further development of TAVI devices but also to improved implantation technologies. Nevertheless, neurological complications are rare but of relevant impact. These are a.e. due to the passage of the TAVI system into an aorta that is often burdened with atheromatous plaques or the necessity to predilate the calcified aortic valve. Studies using cerebral magnetic resonance imaging (MRI) show that the vast majority of patients after TAVI had lesions in the brain that correspond to at least minimal cerebral infarction. Even if these are asymptomatic, various studies have shown that initially asymptomatic infarcts may be associated with an increased incidence of dementia and cognitive impairment, as well as being predictors of later symptomatic infarctions. Changes in hemodynamics after removal of the aortic stenosis could, on the other hand, improve neurocognitive function. Interestingly, the standard methods primarily investigate motor deficits, while neurocognitive function were currently not tested. The influence of a TAVI on the latter functions is therefore unknown. In this study, we aim to differentiate the changes in cognitive functions after a TAVI immediately after the procedure and after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* planned TAVI implantation
* Age ≥ 60
* Intelligence quotient > 80
* Sufficient knowledge of German
* Normal or corrected vision and hearing

Exclusion Criteria:

* Serious neurological or psychiatric diseases that make participation in the trial procedure impossible
* Oncological disease with a life expectancy < 12 months
* pregnancy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is scheduled for TAVI implantation due to symptomatic aortic stenosis. Control is age matched.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-31 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
neurocognitive performance for depression | 6 month post TAVI
  Becks Depression Inventory (BDI)
neurocognitive performance for health status | 6 month post TAVI
  Questionnaire on health status (SF 36)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vorpahl, Prof. Dr., Study Chair — Helios Wuppertal
Locations (1):
- Helios Universitätsklinikum Wuppertal Herzzentrum, Wuppertal, North Rhine-Westphalia, Germany

REFERENCES:
- Available data/document: BECK DEPRESSION INVENTORY — https://www.ismanet.org/doctoryourspirit/pdfs/Beck-Depression-Inventory-BDI.pdf
- Available data/document: SF-36 QUESTIONNAIRE — https://clinmedjournals.org/articles/jmdt/jmdt-2-023-figure-1.pdf